CLINICAL TRIAL: NCT02083016
Title: Ultra-high Density Mapping With Multielectrode Catheter vs Conventional Point by Point Mapping for Ventricular Tachycardia Substrate Ablation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, MD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PentaRay
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Mapping (Other): Both pre and post-ablation mapping will be performed firstly by conventional point by point mapping using a Navistar Thermocool catheter, and secondly by multielectrode contact mapping using a Pentaray catheter. In this group, ablation will be guided by conventional mapping.
  Interventions: Device: Ablation guided by conventional mapping.
- Multielectrode mapping. (Other): Both pre and post-ablation mapping will be performed firstly by multielectrode contact mapping using a Pentaray catheter, and secondly by conventional point by point mapping using a Navistar Thermocool catheter. In this group ablation will be guided by multielectrode contact mapping.
  Interventions: Device: Ablation guided by ultra-high density mapping with multielectrode catheter.

INTERVENTIONS:
Device: Ablation guided by conventional mapping. — Substrate mapping and ablation of ventricular tachycardia.
  Arms: Conventional Mapping
Device: Ablation guided by ultra-high density mapping with multielectrode catheter. — Substrate mapping and ablation of ventricular tachycardia.
  Arms: Multielectrode mapping.

SUMMARY:
Ultra-high density mapping with multielectrode catheter may improve slow conduction channels identification in ventricular tachycardia substrate ablation procedures compared to conventional point by point mapping.

This study compares the ability of both mapping catheters to detect slow conduction channels in areas of myocardial scar and their utility to assess substrate modification after ablation.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled study. Twenty patients with sustained ventricular tachycardia and structurally abnormal ventricle(s) will be prospectively enrolled. In all patients a detailed pre and post-ablation electroanatomical mapping will be performed, and these maps will be merged with CT and/or MRI images. Patients will be randomly assigned to two groups. In Group A patients both pre and post-ablation mapping will be performed firstly by conventional point by point mapping using a Navistar Thermocool catheter, and secondly by multielectrode contact mapping using a Pentaray catheter. In this group, target ablation sites will be guided by point by point map. In Group B patients, both pre and post-ablation mapping will be performed firstly by multielectrode contact mapping using a Pentaray catheter, and secondly by conventional point by point mapping using a Navistar Thermocool catheter. In this group target ablation sites will be guided by multielectrode contact mapping.

Slow conduction channels will be identified by color-coded voltage map adjustment of the lower and upper thresholds and also the presence of fractioned electrograms with the delayed component showing sequential orthodromic activation. The entrances of these channels will be the target of the ablation sites (scar dechanneling technique).

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for ventricular tachycardia substrate ablation.

Exclusion Criteria:

* Pregnant woman.
* Reduced expectancy of life (less than 12 months)
* Patient participating in another clinical study that investigates a drug or device
* Psychologically unstable patient or denies to give informed consent
* Any cause that contraindicate ablation procedure or antiarrhythmic drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mapping and ablation times | During procedure.
  Mapping and ablation times with each mapping system (point by point vs multielectrode mapping).

SECONDARY OUTCOMES:
Scar area correlation with MRI. | Immediately after intervention.
  To assess the correlation between the values of scar area obtained from both electroanatomical mapping systems and those resulting from the analysis of MRI.
Radiofrequency delivery time. | During procedure.
Reduction of residual electrograms with delayed component. | Immediately after intervention.
  Reduction of residual electrograms with delayed component after ablation.
Ventricular tachycardia inducibility after ablation. | Immediately after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Acosta, MD, Principal Investigator — Hospital Clinic of Barcelona; Diego Penela, MD, Principal Investigator — Hosptial Clínic de Barcelona
Locations (1):
- Hospital Clinic Universitari, Barcelona, Barcelona, Spain